CLINICAL TRIAL: NCT05259280
Title: ASPIRE: An Observational Study of the Wellinks Solution Impact on Quality of Life and Clinical Outcomes in Patients With COPD
Brief Title: Observational Study of the Wellinks Solution Impact on Quality of Life and Clinical Outcomes in Patients With COPD
Acronym: ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Convexity Scientific Inc (Industry)
Collaborators: COPD Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WL-2021-02-COPDF
Record Dates: First submitted 2022-01-24; First posted 2022-02-28 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease; Chronic Obstructive Pulmonary Disease Severe; Chronic Obstructive Pulmonary Disease Moderate
Keywords: COPD; Virtual Care; Digital Health; V1C
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Arm 1: Subjects will receive 24 weeks of access to the Wellinks Solution.
  Interventions: Other: Wellinks
- Arm 2 (Experimental): Arm 1: Subjects will receive 24 weeks of access to the Wellinks Solution. The latter 12 weeks will be entirely asynchronous.
  Interventions: Other: Wellinks

INTERVENTIONS:
Other: Wellinks — Digital health and virtual care program for COPD management.

SUMMARY:
The clinical objectives of this study are to determine whether utilization of the Wellinks COPD Solution can improve quality of life for patients with COPD, can reduce healthcare resource utilization over time, and can improve pulmonary function as measured by connected devices.

The nonclinical objectives of this study are to describe the experience of patients using the Wellinks Solution through the assessment of patient engagement with the solution, as well as by patient-reported satisfaction with the solution and their perceived value (e.g., willingness to pay). Qualitative feedback on the features and functionality of the Wellinks Solution will be solicited.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis (confirmed by the patient and assumed based on participation in COPD PPRN)
* Home telephone (landline or mobile) and internet access
* Smartphone: iPhone 6S or later model, running iOS 14.0 or later; Android 6 or later model
* Proficient in English language
* Living/staying in the United States throughout the study duration
* Willing and able to comply with study requirements
* Able to provide written informed consent

Exclusion Criteria:

* Current participation in other interventional clinical trials
* Current participation in a pulmonary rehabilitation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
COPD Symptoms Assessment | Change from baseline to 12 weeks
  Change in self-reported symptoms as collected in the app.
COPD Symptoms Assessment | Change from baseline to 24 weeks
  Change in self-reported symptoms as collected in the app.
COPD Self-Efficacy Scale | Change from baseline to 12 weeks
  Change in COPD Self-Efficacy Scale
COPD Self-Efficacy Scale | Change from baseline to 24 weeks
  Change in COPD Self-Efficacy Scale
Patient-Reported Healthcare Resource Utilization (HRU) | 12 weeks
  Measure of health resource utilization from period baseline to 12 weeks. Emergency room visits. Hospitalizations.
Patient-Reported Healthcare Resource Utilization (HRU) | 24 weeks
  Measure of health resource utilization from period 12 to 24 weeks. Emergency room visits. Hospitalizations.
Modified Medical Research Council Dyspnea Scale (mMRC) | Change from baseline to 12 weeks
  Change in mMRC score. (0-4, 0 is best)
Modified Medical Research Council Dyspnea Scale (mMRC) | Change from baseline to 24 weeks
  Change in mMRC score. (0-4, 0 is best)

OTHER OUTCOMES:
Participant Net Promoter Score (nPS) | 24 weeks
  Measure of the Net Promoter Score - (How likely are you to recommend wellinks to a friend or family member?). Scale: -100 to +100, higher is better.

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen McCreary, Study Director — COPD Foundation
Locations (2):
- United States (2):
  - Wellinks, New Haven, Connecticut
  - COPD Foundation, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pierz KA, Locantore N, McCreary G, Calvey RJ, Hackney N, Doshi P, Linnell J, Sundaramoorthy A, Reed CR, Yates J. Investigation of the Impact of Wellinks on the Quality of Life and Clinical Outcomes in Patients With Chronic Obstructive Pulmonary Disease: Interventional Research Study. JMIR Form Res. 2024 Feb 9;8:e47555. doi: 10.2196/47555. PMID 38335023